CLINICAL TRIAL: NCT01566331
Title: Safe Natural Delivery by Using a New Inflatable Ergonomic Three Chambers Belt
Brief Title: Safe Delivery Using a Belt on the Belly of Pregnant Woman
Acronym: SDB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Erich Cosmi MD, PhD, Director of Maternal and Fetal Medicine, Department of Woman and Child Health, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: unipd
Record Dates: First submitted 2012-03-19; First posted 2012-03-29 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Other Obstetric Trauma - Delivered
Keywords: Safe Delivery; reduction of pain; reduction stage of labor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baby-guardTM (Experimental): Baby-guardTM system, through its ergonomic, three chamber, inflatable abdominal belt, engineered after studies of biomechanics and biophysics, that follows obstetric semiotics, that applies fundal pressure during the second stage of labor in the direction of the pelvic outlet.
  Interventions: Device: Baby-guardTM
- no intervention (No Intervention): Baby-guardTM system, without inflation

INTERVENTIONS:
Device: Baby-guardTM — Baby-guardTM system, through its ergonomic, three chamber, inflatable abdominal belt, engineered after studies of biomechanics and biophysics, that follows obstetric semiotics, that applies fundal pressure during the second stage of labor in the direction of the pelvic outlet, may be of maternal and fetus aid for a safe natural childbirth for their better outcomes
  Other Names: Safety baby guard
  Arms: Baby-guardTM

SUMMARY:
Safety of natural, vaginal labor for parturient, fetus and newborn is one of most important goal among obstetricians, midwifes, scientific society all over the world. Maternal and newborn clinical problems and complications following vaginal delivery cause a big amount of medico-legal problems and high costs in the sanitary field.

Among the maneuvers that are used in the second stage of labor, uterine fundal pressure is one of the most controversial and often diffuse in all over the world, generally not documented, or under reported in medical records . Many Authors affirms that a different new way to push may be of help. This maneuver was introduced by Kristeller, that in 1867 minutely described a procedure to shorten, through the application of a pressure on the uterine fundus whose intensity was quantified by a dynamometer and the duration measured in seconds, the length of the second phase of the labor. Although uterine fundal pressure maneuver was described by Kristeller as the placement of two hands on the uterine fundus and the consequential application of longitudinal steady pressure at a 30- to 45-degree angle directed toward the pelvis, with the avoidance of direct pressure toward the maternal spine, there is no clear definition of the maneuver and no indication for its use has been formally described to date.

The aim of this study was therefore to assess whether the use of the Baby-guardTM system, through its ergonomic, three chamber, inflatable abdominal belt, engineered after studies of biomechanics and biophysics, that follows obstetric semiotics, that applies fundal pressure during the second stage of labor in the direction of the pelvic outlet, may be of maternal and fetus aid for a safe natural childbirth for their better outcomes.

DETAILED DESCRIPTION:
A randomized, single blind, controlled, prospective study was performed. Subjects were nulliparous women who delivered at a community setting hospital (U.O.C. Obstetrics and Gynecology, "San Giuseppe" Hospital, Empoli, Italy) between January 24, 2011 and March 24, 2011. Vaginal deliveries were eligible. Patients were therefore divided into two groups by randomly numbered envelopes upon full dilatation of the cervix, and allocated to the following two groups:

1. The Study Group (n=40 patients) in whom the inflatable belt was applied with the correct pressures (ranging from 80 to 150 mm/Hg, see below the description of the protocol)during Labor and Delivery
2. The Control Group (n=40 women), in whom the belt was inflated with minimal pressures (from 10 to 20 mm/Hg) During Labor and Delivery To test whether differences between experimental groups are statistically significant, the sample-size should be calculated "a priori". To do this, a primary end-point has been identified: incidence of perineal-cervical lacerations. The sample-size (n > 62 subjects for two groups) will be obtained using STATA program by a two-tailed test [alpha level of 0.05 and 90% of statistical power (1-Beta)], to detect statistically significant reduction from 50% to 10% or less with respect the primary end-point. Therefore a randomized sample size of 40 pregnant women per group was chosen to allow for possible refusals or withdrawals.

Data collected from delivery records, retrospectively obtained and reviewed, will include: patient's age, race, parity, patient's body mass index (BMI, kg/m2) at the time of delivery, and body weight change during pregnancy (defined as the difference between maternal pre-pregnant body weight and body weight at delivery), as part of the ante-partum information. For the intra-partum information, gestational age at delivery, duration of second phase of labor, use of intravenous oxytocin, episiotomy, cervical laceration (as requiring surgical repair for hemostasis), severe perineal lacerations (defined as third- or fourth- laceration, while mild perineal laceration was defend as first- or second- perineal laceration), vacuum extraction, forceps delivery, use of uterine fundal pressure maneuver were abstracted. All The study Group will followed up for 15 days after delivery Fetal weight was estimated by the combination of biparietal diameter, abdominal circumference and femur length. The mean percent difference between the predicted and actual weight was 9.6% corresponding to a mean overestimation of 294 g or underestimation of 314 g. These values are consistent with most reports in the literature.

The study will be performed according to the guidelines of the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH); the declaration of Helsinki regarding the Standard operating procedures for clinical investigators (GCP); the General requirements for Clinical investigation of medical devices for human subjects. Finally, the local ethical committee approved the study protocol, and all patients received detailed information about the study and the procedure, to which they gave their written consent.

The inflatable belt (Baby-guardTM ) and study protocol The Baby-guardTM (CABEL s.a.s. Costruzioni Elettroniche, Pistoia, Italy) consists of a disposable, ergonomic, three chambers, inflatable belt, and a detector of electro-physiological signals from maternal abdomen (i.e. fetal heart and maternal heart signals - Figure 1). myographic uterine activity). Three chambers that can be separately swollen one from the other in order to repositioning fetal body compose the inflatable belt. The three belt chambers are filled according to the pressures set by the operator (midwife/MD) and allow to gently positioning of the fetus in the wright position towards the pelvis. Once the correct fetal position has been obtained, all three chambers are inflated in synchronously with uterine contraction. The maternal and fetal monitoring unit is composed by a touch-screen computer, that records electro-physiological signals collected by a signal amplifier deriving from the mother (uterine contractions and the maternal heart rate) and the fetus (fetal heart rate and the possibility of Doppler parameters of fetal heart). All parameters and signals detected by the Baby-guardTM system are storable on the touch-screen computer hard disk, as per request of the European Community rules on safety (UNI EN60601)].

This study reports only the part regarding results and outcomes of parturient and neonates.

At the beginning of the uterine contraction, as referred by the patients and revealed by the electro-physiological signals recorded, the midwife/MD, if necessary, inflated 30-50 mmHg of air pressure into the lateral chambers of the inflatable belt to correctly align the fetus avoiding his malpositioning with respect to the pelvis. After monitoring the duration of spontaneous uterine contractions, the midwife/MD therefore inflated from 80 to 150 mm/Hg (for the Study Group) or from 10 to 20 mm/Hg (for the Control Group) of air into the ergonomic belt for 30 sec. Fundal pressure was applied at a 30-40° angle to the spine in the direction of the pelvic outlet through the inflatable belt, standardizing the force and surface area of application (980 cm2). The frequency of inflation was limited to fewer than 6 times per 20 min. followed by a pause of 10 min. All the women, whether randomized to the Study or the Control group, received standard management of the second stage of labor, which includes one-to-one support, fetal heart rate monitoring, and care from midwife. Operative deliveries were performed if clinically indicated. As a uterine contraction started, the inflatable obstetric belt was inflated synchronously and maintained at the pressure above indicated for 30 sec. by the midwife/MD. The Baby-guardTM was not used for more than 2 hours till delivery. The obstetrician, the midwife and the patients were blind to whether the belt was inflated with sufficient pressure (from 80 to 150 mm/Hg for the Study Group) or not (from 10 to 20 mm/Hg for the Control Group).

Outcomes of the study Outcome measures in this study were the perineal and cervical lacerations incidence, the use of uterine fundal pressure maneuver (Kristeller manouvre), the incidence of vacuum extractions, cesarean section incidence during labor, second stage of labor duration; maternal psychological and physical fatigue, maternal request of cesarean section during labor, and absence of neonatal intensive care unit admissions.

At the time of discharge to home, patients' satisfaction with the inflatable belt was evaluated asking them to score about the degree of psychological and physical fatigue with the Baby-guardTM by marking a 10-cm visual analogue scale (VAS) from 0 (minimal) to 10 (optimal). Patients were also asked about the usefulness of the inflatable belt assistance to delivery. The number of cesarean section requests during the second phase of labor was also evaluated.

Statistical analysis All data were analyzed with the STATA software (StataCorp LP, College Station, Texas, USA), and were expressed as mean ± SD (range) or as number (%) of cases. Comparisons of proportions and means between groups (study vs control) were done using the χ2 test (or Fisher exact test, if suitable) and, independent t-test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* women in active labor at term in primipara with maternal age ranging from 23 to 42 years, with a singleton fetus in vertex presentation.
* the onset of second stage was defined as full dilatation of the cervix identified by digital examination

Exclusion Criteria:

* preterm labor (gestational age below 37 weeks)
* breech or transverse presentation
* suspected fetal macrosomia
* gestational diabetes
* pregnancy-induced hypertension
* abnormalities of placentation (low lying placenta, abruptio placenta)
* uterine structural abnormalities
* history of previous uterine scar
* fetal heart rate abnormalities at the time of enrollment (bradycardia, tachycardia or prolonged variable decelerations).

Ages: 23 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: luisa Acanfora, MD, Study Chair — University of Florence
Locations (1):
- University of Padua, Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoogsteder PH, Pijnenborg JM. Use of uterine fundal pressure maneuver at vaginal delivery and risk of severe perineal laceration. Arch Gynecol Obstet. 2010 Mar;281(3):579-80. doi: 10.1007/s00404-009-1229-3. Epub 2009 Sep 23. No abstract available. PMID 19774390
- [Background] Cosner KR. Use of fundal pressure during second-stage labor. A pilot Study. J Nurse Midwifery. 1996 Jul-Aug;41(4):334-7. doi: 10.1016/0091-2182(96)00033-x. PMID 8828318
- [Background] Api O, Api M. Uterine fundal pressure and duration of the second stage of labor: A randomized controlled trial. Acta Obstet Gynecol Scand. 2009;88(11):1297-8. doi: 10.3109/00016340903214999. No abstract available. PMID 19900147
- [Derived] Acanfora L, Rampon M, Filippeschi M, Marchi M, Montisci M, Viel G, Cosmi E. An inflatable ergonomic 3-chamber fundal pressure belt to assist vaginal delivery. Int J Gynaecol Obstet. 2013 Jan;120(1):78-81. doi: 10.1016/j.ijgo.2012.07.025. Epub 2012 Oct 16. PMID 23083494

RESULTS

PARTICIPANT FLOW:
Groups:
- Baby-guardTM Minimal Inflation: Baby-guardTM with minimal inflation who expected natural delivery
Period: Overall Study
Arm/Group | Baby-guardTM | Baby-guardTM Minimal Inflation
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baby-guardTM With Minimal Inflation: Baby-guardTM system, with minimal inflation in women who expected natural delivery
- Total: Total of all reporting groups
Arm/Group | Baby-guardTM | Baby-guardTM With Minimal Inflation | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.97 (5.16) | 31.45 (1.2) | 31.1 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Partecipant With Perineal Laceration
Description: The following types of lacerations were recorded during delivery: cervical laceration; mild perineal lacerations (defined as 1-2 lacerations); severe perineal lacerations (defined as 3-4 lacerations)
Time Frame: after delivery
Population: intervention in normal pregnancies at term during labor and delivery
Measure: Number; unit: participants
Arm/Group | Baby Belt Device Group | Baby-guardTM With Minimal Inflation
Number analyzed (Participants) | 40 | 40
participants | 3 | 31

ADVERSE EVENTS:
Time Frame: discomfort during labor
Groups:
- Baby Birth: group delivering with baby birth
- Baby Birth With Minimal Inflation: group delivering with dwvice and minimal inflation
Arm/Group | Baby Birth | Baby Birth With Minimal Inflation
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No